CLINICAL TRIAL: NCT06536855
Title: Faster Elimination of HPV Infection and Cervical Cancer Using Concomitant HPV Vaccination and HPV Screening: A Demonstration Project in Rwanda
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rwanda Biomedical Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Karolinska Institutet (Other); Center for Family Health Research/Projet San Francisco (Unknown); ELEKTA Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FasterHPV01
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Intervention Model Description: At the first visit we will administer Gardasil 9 to women aged 23 to 29 years and screening them for HPV to get baseline information, after 24 months at the second visit, provide the second dose and screen again for HPV to be able to compare HPV prevalence at baseline and 24 months after administering the second dose of vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gardasil 9 Arm (Experimental): The study is open label with only one arm that will receive the vaccine
  Interventions: Biological: Gardasil 9

INTERVENTIONS:
Biological: Gardasil 9 — GARDASIL 9 is a vaccine indicated in females 9 through 45 years of age for the prevention of cervical, vulvar, vaginal, anal, oropharyngeal and other head and neck cancers caused by human papillomavirus (HPV) Types 16, 18, 31, 33, 45, 52, and 58; cervical, vulvar, vaginal, and anal precancerous or dysplastic lesions caused by HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58; and genital warts caused by HPV Types 6 and 11.
  GARDASIL 9 is indicated in males 9 through 45 years of age for the prevention of anal, oropharyngeal and other head and neck cancers caused by HPV Types 16, 18, 31, 33, 45, 52, and 58; anal precancerous or dysplastic lesions caused by HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58; and genital warts caused by HPV Types 6 and 11.
  Other Names: HPV/DNA testing (Gynotyping)

SUMMARY:
Cervical cancer is the fourth most frequently diagnosed cancer and the fourth leading cause of cancer death in women, with an estimated 604,000 new cases and 342,000 deaths worldwide in 2020. Rwanda is among countries with a high burden cervical cancer, with an annual incidence of 28.2/100,000 women (1,229 new cases in 2020) and a mortality rate of 20.1/100,000 (829 deaths in 2018) according to WHO (IARC 2020).

Cervical cancer is almost completely preventable because of the highly effective primary (HPV vaccine) and secondary (HPV screening) prevention measures. However, these measures have not been equitably implemented across and within LMICs countries.

Given the current situation, where the screening coverage is still low due to financial and operational challenges, it will take many years to achieve the elimination targets as included in the global elimination strategy. We are proposing to implement an innovative strategy to accelerate the elimination of cervical cancer in Rwanda consisting of concomitant HPV vaccination and HPV screening for young women aged 23-29 years old.

HPV screening and vaccination are complementary preventive options often implemented as separate public health programs. This project proposal aims to address this disconnect by combining both strategies with the ultimate purpose of accelerating the reduction of cervical cancer incidence and mortality in Rwanda and making the programs both cost-effective and sustainable.

Primary objective

The study aims to evaluate whether organized, concomitant HPV vaccination and HPV screening offered to girls and women aged 23-29 years will result in more rapid elimination of HPV infections in the target districts in Rwanda.

The study design is a before-after study design of the intervention, where the projected incidences and prevalence at the 2-year follow-up visit are modeled using the data from the baseline visit, with evaluation using Observed/expected numbers.

Secondary objectives

The study will evaluate whether concomitant vaccination and cervical screening result in an improved efficiency and/or safety of the cervical cancer screening program. These objectives will be examined among women who participated in the combined screening and vaccination study.

i) Protection of Gardasil 9 against HPV infection and against CIN2+ by Gardasil 9 HPV vaccine types in 23 to 29-year-old women from the study districts. This analysis will be performed every 2 years, and the first analysis will determine the effectiveness of one-dose vaccination (incident infections of HPV vaccine types at 2 years), whereas all subsequent analysis will determine the effect of 2-dose vaccinations. The study will be powered to detect a decline in invasive cervical cancer among the study participants, using the cervical cancer incidence in the surrounding districts of Rwanda as the reference.

ii) Efficiency will also be measured by the yield of histopathologically confirmed high-grade cervical cancer precursors or cancer (cervical intraepithelial neoplasia grade 2, 3, or cervical cancer) in relation to the consumption of resources and convenience for the women, using the yield at the baseline visit (10% of women tested) as the comparator. The hypothesis is that 2 years after vaccination, there will be only a few incident infections (only some old, persistent infections) resulting in high PPV and high yield of CIN2+ at modest consumption of resources.

End of the study

One screening interval (2 years) after the last visit of the last subject, defined as the day the last study subject receives her second vaccination.

The study will be implemented in 4 districts of Rwanda covering 100,000 women aged 23 to 29 years old. We will use Gardasil 9, the HPV the second generation HPV Vaccine manufactured by Merck.

ELIGIBILITY:
Inclusion Criteria:

Eligible women will include women within the age range of 23-29, who have not opted out of the screening program and who consent to participate in the study

Exclusion Criteria:

* Known history of severe allergic reaction or hypersensitivity to any of the components of the HPV vaccine. (For GARDASIL 9: Amorphous aluminium hydroxyphosphate sulphate adjuvant, Sodium chloride, L-histidine, Polysorbate 80, or Sodium borate)
* Known history of immune-related disorders
* Current acute severe febrile illness, except for minor infections such as a cold, mild upper respiratory infection, or low-grade fever.
* Administration of immunoglobulin or blood-derived products within 6 months prior to the scheduled HPV vaccine first dose
* Current pregnancy (reported)
* Women with a total hysterectomy

Ages: 23 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females are the only ones concerned by Cervical cancer
Enrollment: 100000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV infections in the study participants | 24 months
  To evaluate whether organised, concomitant HPV vaccination and HPV screening offered to women aged 23-29 will result in faster elimination of HPV infection in the study districts in Rwanda, using before-design modeling the expected numbers after the intervention.
  Overall and type-specific prevalence and incidence of HPV will be obtained from the HPV screening at 2 years. Observed numbers will be compared to the predicted (expected numbers).

SECONDARY OUTCOMES:
Prevalence of histopathologically confirmed high-grade cervical cancer precursors or cancer (cervical intraepithelial neoplasia grade 2, 3, or cervical cancer) (CIN2+) by HPV type in the lesion. | 24 months
  The study screenings will determine the prevalence of high-grade cervical cancer precursors or cancer (cervical intraepithelial neoplasia grade 2, 3, or cervical cancer) (CIN2+) by HPV type in the lesion at baseline and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Uwinkindi, MD, Msc Epi, Principal Investigator — Rwanda Biomedical Centre; Claude Mambo Muvunyi, MD, PhD, Study Chair — Rwanda Biomedical Centre; Joachim Dillner, MD, PhD, Study Director — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
We plan to share aggregated results. The IPD will not be shared and this is in line with Rwanda National Ethics Committee and GCP principles

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Bosch FX, Lorincz A, Munoz N, Meijer CJ, Shah KV. The causal relation between human papillomavirus and cervical cancer. J Clin Pathol. 2002 Apr;55(4):244-65. doi: 10.1136/jcp.55.4.244. PMID 11919208
- [Result] Guan P, Howell-Jones R, Li N, Bruni L, de Sanjose S, Franceschi S, Clifford GM. Human papillomavirus types in 115,789 HPV-positive women: a meta-analysis from cervical infection to cancer. Int J Cancer. 2012 Nov 15;131(10):2349-59. doi: 10.1002/ijc.27485. Epub 2012 Mar 20. PMID 22323075
- [Result] Denny L, Adewole I, Anorlu R, Dreyer G, Moodley M, Smith T, Snyman L, Wiredu E, Molijn A, Quint W, Ramakrishnan G, Schmidt J. Human papillomavirus prevalence and type distribution in invasive cervical cancer in sub-Saharan Africa. Int J Cancer. 2014 Mar 15;134(6):1389-98. doi: 10.1002/ijc.28425. Epub 2013 Nov 14. PMID 23929250
- [Result] Carrillo-Garcia A, Ponce-de-Leon-Rosales S, Cantu-de-Leon D, Fragoso-Ontiveros V, Martinez-Ramirez I, Orozco-Colin A, Mohar A, Lizano M. Impact of human papillomavirus coinfections on the risk of high-grade squamous intraepithelial lesion and cervical cancer. Gynecol Oncol. 2014 Sep;134(3):534-9. doi: 10.1016/j.ygyno.2014.06.018. Epub 2014 Jun 27. PMID 24979052
- [Result] Cheng L, Wang Y, Du J. Human Papillomavirus Vaccines: An Updated Review. Vaccines (Basel). 2020 Jul 16;8(3):391. doi: 10.3390/vaccines8030391. PMID 32708759
- [Result] Ronco G, Dillner J, Elfstrom KM, Tunesi S, Snijders PJ, Arbyn M, Kitchener H, Segnan N, Gilham C, Giorgi-Rossi P, Berkhof J, Peto J, Meijer CJ; International HPV screening working group. Efficacy of HPV-based screening for prevention of invasive cervical cancer: follow-up of four European randomised controlled trials. Lancet. 2014 Feb 8;383(9916):524-32. doi: 10.1016/S0140-6736(13)62218-7. Epub 2013 Nov 3. PMID 24192252
- [Result] Knaul FM, Farmer PE, Krakauer EL, De Lima L, Bhadelia A, Jiang Kwete X, Arreola-Ornelas H, Gomez-Dantes O, Rodriguez NM, Alleyne GAO, Connor SR, Hunter DJ, Lohman D, Radbruch L, Del Rocio Saenz Madrigal M, Atun R, Foley KM, Frenk J, Jamison DT, Rajagopal MR; Lancet Commission on Palliative Care and Pain Relief Study Group. Alleviating the access abyss in palliative care and pain relief-an imperative of universal health coverage: the Lancet Commission report. Lancet. 2018 Apr 7;391(10128):1391-1454. doi: 10.1016/S0140-6736(17)32513-8. Epub 2017 Oct 12. No abstract available. PMID 29032993
- [Result] Binagwaho A, Wagner CM, Gatera M, Karema C, Nutt CT, Ngabo F. Achieving high coverage in Rwanda's national human papillomavirus vaccination programme. Bull World Health Organ. 2012 Aug 1;90(8):623-8. doi: 10.2471/BLT.11.097253. Epub 2012 May 23. PMID 22893746
- [Result] Gatera M, Bhatt S, Ngabo F, Utamuliza M, Sibomana H, Karema C, Mugeni C, Nutt CT, Nsanzimana S, Wagner CM, Binagwaho A. Successive introduction of four new vaccines in Rwanda: High coverage and rapid scale up of Rwanda's expanded immunization program from 2009 to 2013. Vaccine. 2016 Jun 17;34(29):3420-6. doi: 10.1016/j.vaccine.2015.11.076. Epub 2015 Dec 17. PMID 26704259
- [Result] Schiller JT, Castellsague X, Garland SM. A review of clinical trials of human papillomavirus prophylactic vaccines. Vaccine. 2012 Nov 20;30 Suppl 5(0 5):F123-38. doi: 10.1016/j.vaccine.2012.04.108. PMID 23199956
- [Result] Bogaards JA, Coupe VM, Meijer CJ, Berkhof J. The clinical benefit and cost-effectiveness of human papillomavirus vaccination for adult women in the Netherlands. Vaccine. 2011 Nov 8;29(48):8929-36. doi: 10.1016/j.vaccine.2011.09.055. Epub 2011 Sep 22. PMID 21945961
- [Result] Lei J, Ploner A, Elfstrom KM, Wang J, Roth A, Fang F, Sundstrom K, Dillner J, Sparen P. HPV Vaccination and the Risk of Invasive Cervical Cancer. N Engl J Med. 2020 Oct 1;383(14):1340-1348. doi: 10.1056/NEJMoa1917338. PMID 32997908
- [Result] Karimi-Zarchi M, Allahqoli L, Nehmati A, Kashi AM, Taghipour-Zahir S, Alkatout I. Can the prophylactic quadrivalent HPV vaccine be used as a therapeutic agent in women with CIN? A randomized trial. BMC Public Health. 2020 Feb 27;20(1):274. doi: 10.1186/s12889-020-8371-z. PMID 32106837
- [Result] Castellsague X, Munoz N, Pitisuttithum P, Ferris D, Monsonego J, Ault K, Luna J, Myers E, Mallary S, Bautista OM, Bryan J, Vuocolo S, Haupt RM, Saah A. End-of-study safety, immunogenicity, and efficacy of quadrivalent HPV (types 6, 11, 16, 18) recombinant vaccine in adult women 24-45 years of age. Br J Cancer. 2011 Jun 28;105(1):28-37. doi: 10.1038/bjc.2011.185. Epub 2011 May 31. PMID 21629249
- [Result] Skinner SR, Szarewski A, Romanowski B, Garland SM, Lazcano-Ponce E, Salmeron J, Del Rosario-Raymundo MR, Verheijen RH, Quek SC, da Silva DP, Kitchener H, Fong KL, Bouchard C, Money DM, Ilancheran A, Cruickshank ME, Levin MJ, Chatterjee A, Stapleton JT, Martens M, Quint W, David MP, Meric D, Hardt K, Descamps D, Geeraerts B, Struyf F, Dubin G; VIVIANE Study Group. Efficacy, safety, and immunogenicity of the human papillomavirus 16/18 AS04-adjuvanted vaccine in women older than 25 years: 4-year interim follow-up of the phase 3, double-blind, randomised controlled VIVIANE study. Lancet. 2014 Dec 20;384(9961):2213-27. doi: 10.1016/S0140-6736(14)60920-X. Epub 2014 Sep 1. PMID 25189358
- [Result] Ibrahim Khalil A, Zhang L, Muwonge R, Sauvaget C, Basu P. Efficacy and safety of therapeutic HPV vaccines to treat CIN 2/CIN 3 lesions: a systematic review and meta-analysis of phase II/III clinical trials. BMJ Open. 2023 Oct 24;13(10):e069616. doi: 10.1136/bmjopen-2022-069616. PMID 37879679
- [Result] Sayinzoga F, Umulisa MC, Sibomana H, Tenet V, Baussano I, Clifford GM. Human papillomavirus vaccine coverage in Rwanda: A population-level analysis by birth cohort. Vaccine. 2020 May 19;38(24):4001-4005. doi: 10.1016/j.vaccine.2020.04.021. Epub 2020 Apr 24. PMID 32336599
- [Result] Lehtinen M, Baussano I, Paavonen J, Vanska S, Dillner J. Eradication of human papillomavirus and elimination of HPV-related diseases - scientific basis for global public health policies. Expert Rev Vaccines. 2019 Feb;18(2):153-160. doi: 10.1080/14760584.2019.1568876. Epub 2019 Feb 7. PMID 30657348
- See also: Globocan estimate, Rwanda 2020 — https://gco.iarc.fr/today/data/factsheets/populations/646-rwanda-fact-sheets.pdf
- See also: IARC Monographs on the Evaluation of Carcinogenic Risks to Humans Volume 90 — https://publications.iarc.fr/Book-And-Report-Series/Iarc-Monographs-On-The-Identification-Of-Carcinogenic-Hazards-To-Humans/Human-Papillomaviruses-2007
- See also: WHO guideline for screening and treatment of cervical precancer lesions for cervical cancer prevention — https://www.who.int/publications/i/item/9789240030824
- See also: Global strategy to accelerate the elimination of cervical cancer as a public health problem — https://www.who.int/publications/i/item/9789240014107
- See also: Human papillomavirus vaccines: WHO position paper (2022 update) — https://apps.who.int/iris/bitstream/handle/10665/365351/WER9750-645-672-engfre.pdf?sequence=1&isAllowed=y.